CLINICAL TRIAL: NCT06118840
Title: Assessing the Impact of an Artificial Intelligence-Based Model for Intracranial Aneurysm Detection in CT Angiography on Patients' Diagnosis and Outcomes: The IDEAL Study - A Web-Based Multicenter, Double-Blinded Randomized Controlled Trial
Brief Title: IDEAL Study: Blinded RCT for the Impact of AI Model for Cerebral Aneurysms Detection on Patients' Diagnosis and Outcomes
Acronym: IDEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang longjiang,MD, Head of Radiology, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2022NZKY-015-05
Record Dates: First submitted 2022-08-29; First posted 2023-11-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Aneurysm; CT Angiography; Deep Learning; Double Bind Interaction
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants, nurses acquiring for patients' consent and radiographers acquiring head computered tomograhy angiography exams will be blinded to the randomization as it is automatically performed after the exam has been acquired.
  A Sham-AI for the automatic detection of intracranial aneurysms has been delicately designed to mimic the True-AI model with a sensitivity close to zero and a similar specificity to True-AI. Thereforem, the participating radiologists interpreting head computered tomograhy angiography exams will also be blinded to the allocation of the AI models.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True-AI-integrated intracranial aneurysms diagnosis strategy (Experimental): For patients who underwent head CTA and assigned to True-AI group, they will be diagnosed by a radiologist who are aided by the True-AI-integrated intracranial aneurysms diagnosis strategy.
  Interventions: Device: True-AI-integrated intracranial aneurysms diagnosis strategy
- Sham-AI-integrated intracranial aneurysms diagnosis strategy (Sham Comparator): For patients who underwent head CTA and assigned to Sham-AI group, they will be diagnosed by a radiologist who are aided by the Sham-AI-integrated intracranial aneurysms diagnosis strategy. To mimic the True-AI, the Sham-AI had a sensitivity close to 0% and a similar specificity to the True-AI.
  Interventions: Device: Sham-AI-integrated intracranial aneurysms diagnosis strategy

INTERVENTIONS:
Device: True-AI-integrated intracranial aneurysms diagnosis strategy — The True-AI deep-learning based model for intracranial aneurysms detection had a patient-wise sensitivity, lesion-wise sensitivity and specificity of 0.96, 0.87, and 0.80 in the internal validation dataset.
  Arms: True-AI-integrated intracranial aneurysms diagnosis strategy
Device: Sham-AI-integrated intracranial aneurysms diagnosis strategy — The Sham-AI deep-learning based model for intracranial aneurysms detection is designed to have a sensitivity close to 0% and a similar specificity to the True-AI. In the internal validation dataset, the Sham-AI had a patient-wise sensitivity, lesion-wise sensitivity, specificity of 0.02, 0.01, and 0.80, respectively.
  Arms: Sham-AI-integrated intracranial aneurysms diagnosis strategy

SUMMARY:
This study (IEDAL study) intends to prospectively enroll more than 6450 patients who will undergo head CT angiography (CTA) scanning in the outpatient clinic. It will be carried out in 21 hospitals in more than 10 provinces in China. The patient's head CTA images will be randomly assigned to the True-AI and Sham-AI group with a ratio of 1:1, and the patients and radiologists are unaware of the allocation. The primary outcomes are sensitivity and specificity of detecting intracranial aneurysms. The secondary outcomes focus on the prognosis and outcomes of the patients.

DETAILED DESCRIPTION:
A multicenter, prospective, double-blind, randomized controlled trial will be conducted (IDEAL study). Patients who are scheduled to undergo cranial CT angiography (CTA) scanning will be randomly divided into two groups with a ratio of 1:1, one of the group will be assigned to True-AI aided intracranial aneurysms diagnosis strategy (True-AI group) and the other will be assigned to Sham-AI aided intracranial aneurysms diagnosis strategy (Sham-AI group, which has a sensitivity close to 0% and a similar specificity to True-AI). The primary outcomes are diagnostic sensitivity and specificity of detecting aneurysms. Secondary endpoints include other diagnostic performance indexes for intracranial aneurysms; diagnostic performances for other intracranial lesions for intracranial arterial stenosis, occlusion, and intracranial tumors; detection rates of intracranial lesions according to Radiology Reports; workload of head CTA interpretation; resource use; treatment-related indexes during patient follow-up (e.g. clinical follow-up, hospitalization, rate of patients undergoing DSA); life quality; outcomes of aneurysm-related events; repeat head CTA or MRA at 12-month follow; cost-effectiveness analysis between intervention and control arm to evaluate the short- and longterm influence of AI system to the routine practice and patients' prognosis and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients and outpatients who are scheduled for head CTA scanning.

Exclusion Criteria:

* Age under 18 years.
* Patients with contraindications to CTA.
* Modified Rankin Scale (mRS) score > 3.
* Refuse to sign informed consent.
* Participation in other clinical studies of intracranial aneurysms.
* Patients with failed head CTA scanning or incomplete image data, or poor image quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6450 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To compare diagnostic sensitivity of intracrnial aneurysms between intervention and control arm. | 6 months.
  The proportion of examinations in which at least one aneurysm is discovered and indicated among groundtruth aneurysms.
To compare diagnostic specificity of intracrnial aneurysms between intervention and control arm. | 6 months.
  The proportion of examinations in which no aneurysms are spotted by the reader among groundtruth non-aneurysms.

SECONDARY OUTCOMES:
To compare other diagnostic performances for intracranial aneurysms between intervention and control arm. | 6 months.
  To compare accuracy, lesion-wise sensitivity, positive predictive value and negative predictive value for intracranial aneurysms between intervention and control arm.
To compare diagnostic performances for other intracranial lesions between intervention and control arm. | 6 months.
  The sensitivity, specificity, accuracy, positive predictive value and negative predictive value for intracranial arterial stenosis, occlusion, and intracranial tumors are compared between intervention and control arm.
To compare detection rates of intracranial lesions according to Radiology Reports between intervention and control arm. | 6 months.
  Detection rates of intracranial aneurysms, intracranial arterial stenosis, occlusion, and intracranial tumors according to Radiology Reports are compared between intervention and control arm.
To assess the workload of head CT angiography interpretation. | 6 months.
  Time of interpreting head CT angiography images, number of consensus meeting are compared between intervention and control arm.
To assess resource use. | At 3-month and 12-month follow-up.
  The number of care encounters (in-person) during follow-up, total number of outpatient encounters for aneurysm referral, total number of cerebral artery disease testing are compared between intervention and control arm.
Rate of patients of subsequent hospitalization during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of patients of subsequent hospitalization is compared between intervention and control arm.
In-hospital mortality rate during patient follow-up. | At 3-month and 12-month follow-up.
  In-hospital mortality rate is compared between intervention and control arm.
Morbidity (modified Rankin Score ≥ 3) from intracranial haemorrhage or treatment during patient follow-up. | At 3-month and 12-month follow-up.
  Morbidity (modified Rankin Score ≥ 3) from intracranial haemorrhage or treatment is compared between intervention and control arm.
Length of hospital stay during patient follow-up. | At 3-month and 12-month follow-up.
  Length of hospital stay is compared between intervention and control arm.
Rate of hospitalization for intracranial aneurysms during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of hospitalization for intracranial aneurysms is compared between intervention and control arm.
Rate of patients undergoing digital subtraction angiography (DSA) during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of patients undergoing digital subtraction angiography (DSA) is compared between intervention and control arm.
Detection rate of intracranial aneurysms among digital subtraction angiographys (DSA) during patient follow-up. | At 3-month and 12-month follow-up.
  Detection rate of intracranial aneurysms among digital subtraction angiographys (DSA) is compared between intervention and control arm.
Detection rate of no abnormality among digital subtraction angiographys (DSA) during patient follow-up. | At 3-month and 12-month follow-up.
  Detection rate of no abnormality among digital subtraction angiographys (DSA) is compared between intervention and control arm.
Distribution of the methods for aneurysms management (conservative/coil/clip/others) during patient follow-up. | At 3-month and 12-month follow-up.
  Distribution of the methods for aneurysms management (conservative/coil/clip/others) is compared between intervention and control arm.
Rates of aneurysm treatment related complications during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of aneurysm treatment related complications (intraoperative rupture, stroke, et al) is compared between intervention and control arm.
Rate of recurrence or residual of intracranial aneurysm after surgery during patient follow-up. | At 12-month follow-up.
  Rate of recurrence or residual of intracranial aneurysm after surgery is compared between intervention and control arm.
Life quality assessed by EuroQol 5-Dimensional, 5-Level (EQ-5D-5L) during patient follow-up. | At 3-month and 12-month follow-up.
  Life quality assessed by EuroQol 5-Dimensional, 5-Level (EQ-5D-5L) scores are compared between intervention and control arm, which ranges from 5 to 25, and higher scores mean a worse outcome.
Restrictions in daily activities assessed by Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P) scores during patient follow-up. | At 3-month and 12-month follow-up.
  Restrictions in daily activities assessed by Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P) scores are compared between intervention and control arm.
Sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) during patient follow-up. | At 3-month and 12-month follow-up.
  Sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) is compared between intervention and control arm, which ranges from 0 to 21, and higher scores mean a worse outcome.
Depression Screening assessed by Patient Health Questionnaire-9 (PHQ-9) scores during patient follow-up. | At 3-month and 12-month follow-up.
  Depression Screening assessed by Patient Health Questionnaire-9 (PHQ-9) scores are compared between intervention and control arm, which ranges from 0 to 27, and higher scores mean a worse outcome.
Anxiety and depression assessed by Hospital Anxiety and Depression Scale (HADS) scores during patient follow-up. | At 3-month and 12-month follow-up.
  Anxiety and depression assessed by Hospital Anxiety and Depression Scale (HADS) scores are compared between intervention and control arm, which ranges from 0 to 21, and higher scores mean a worse outcome.
General health assessed by Short-Form 36 Health Survey (SF-36) scores during patient follow-up. | At 3-month and 12-month follow-up.
  General health assessed by Short-Form 36 Health Survey (SF-36) scores are compared between intervention and control arm.
Functional outcome assessed by Modified Rankin Scale (mRS) scores during patient follow-up. | At 3-month and 12-month follow-up.
  Functional outcome assessed by Modified Rankin Scale (mRS) scores are compared between intervention and control arm, which ranges from 0 to 5, and higher scores mean a worse outcome.
All-cause mortality during patient follow-up. | At 3-month and 12-month follow-up.
  All-cause mortality is compared between intervention and control arm.
Rate of aneurysm growth during patient follow-up. | At 12-month follow-up.
  Rate of aneurysm growth is compared between intervention and control arm.
Rate of aneurysm rupture during patient follow-up. | At 12-month follow-up.
  Rate of aneurysm rupture is compared between intervention and control arm.
Rate of subarachnoid hemorrhage (SAH) during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of subarachnoid hemorrhage (SAH) is compared between intervention and control arm.
Rate of other types of stroke (hemorrhagic stroke, ischemic stroke) during patient follow-up. | At 3-month and 12-month follow-up.
  Rate of other types of stroke (hemorrhagic stroke, ischemic stroke) is compared between intervention and control arm.
Mortality of aneurysms-rupture during patient follow-up. | At 3-month and 12-month follow-up.
  Mortality of aneurysms-rupture is compared between intervention and control arm.
Morphological change by head CTA or magnetic resonance angiography at the 12-month follow-up. | At 12-month follow-up.
  Morphological change by head CTA or magnetic resonance angiography is assessed.

OTHER OUTCOMES:
Patient-wise sensitivity and specificity at different centers, provinces, geography areas and levels of physician. | 6 months.
  To compare diagnostic performances of patient-wise sensitivity and specificity for intracranial aneurysms between intervention and control arm in subgroups of different centers, provinces, geography areas and physician level.
Subgroup analysis of different size (< 5 mm vs. ≥ 5 mm), locations of intracranial aneurysms. | 6 months.
  To compare diagnostic performances for intracranial aneurysms between intervention and control arm in subgroups of different size (internal carotid artery vs. middle cerebral artery vs. anterior cerebral artery vs. posterior communication artery vs. anterior communication artery vs. vertebral basilar artery vs. others), locations (internal carotid artery vs. middle cerebral artery vs. anterior cerebral artery vs. posterior communication artery vs. anterior communication artery vs. vertebral basilar artery vs. others) of intracranial aneurysms.
Subgroup analysis of different gender (male vs. female), age (≤ 54 years or. >54 years), subarachnoid hemorrhage status (with vs. without SAH) of patients | 6 months.
  To compare diagnostic performances for intracranial aneurysms between intervention and control arm in subgroups of different gender (male vs. female), age (≤ 54 years or. >54 years), subarachnoid hemorrhage status (with vs. without SAH) of patients.
Patient-wise sensitivity and specificity for patients with previous head digital subtraction angiography or surgery or not. | 6 months.
  To compare diagnostic performances of patient-wise sensitivity and specificity for intracranial aneurysms between intervention and control arm in subgroups of patients with previous head angiography or surgery or not.
Patient-wise sensitivity and specificity for patients with subsequent head digital subtraction angiography or surgery or not. | 6 months.
  To compare diagnostic performances of patient-wise sensitivity and specificity for intracranial aneurysms between intervention and control arm in subgroups of patients with subsequent head angiography or surgery or not.
Ethical safety outcomes. | 6 months.
  The monthly reported detection rates of intracranial aneurysms, tumors, stenosis, and occlusive are calculated and compared with the reported detection rates in the previous 3 months during the trial.
Learning curve of AI-augmented intracranial aneurysm diagnosis. | 6 months.
  Dynamic changes in sensitivity and specificity of aneurysm diagnosis from the first 7-days through to the last 7-days of all center trials.

CONTACTS AND LOCATIONS:
Overall Officials: Trial Manager, Principal Investigator — Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (21):
- China (21):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shiyan People's Hospital, Shiyan, Hubei
  - Research Institute Of Medical Imaging Jinling Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Yidu Central Hospital Affiliated to Shandong Second Medical University, Weifang, Shandong
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hainan General Hospital, Haikou
  - The First People's Hospital of Kashgar Region, Kashgar
  - University Second Hospital, Lanzhou
  - First People's Hospital of Lianyungang, Lianyungang
  - Ma'anshan People's Hospital, Ma’anshan
  - BenQ Medical Center, Affiliated BenQ Hospital of Medical School, Nanjing Medical University, Nanjing
  - Long Gang Central Hospital of Shenzhen, Shenzhen
  - The Affiliated Suqian First Hospital of Nanjing Medical University, Suqian
  - Tianjin Medical University General Hospital, Tianjin
  - General Hospital of Ningxia Medical University, Yinchuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Z, Hu B, Lu M, Chen Z, Zhang M, Yu Y, Zhou C, Zhong J, Wu B, Zhang X, Wei Y, Zhang LJ; China Aneurysm AI Project Group. Assessing the Impact of an Artificial Intelligence-Based Model for Intracranial Aneurysm Detection in CT Angiography on Patient Diagnosis and Outcomes (IDEAL Study)-a protocol for a multicenter, double-blinded randomized controlled trial. Trials. 2024 Jun 4;25(1):358. doi: 10.1186/s13063-024-08184-9. PMID 38835091